CLINICAL TRIAL: NCT04784884
Title: Pilot Study of Intraoperative Tissue Differentiation and Vascular Perfusion Using Intraoperative Hyperspectral Imaging (HSI) in Benign and Malignant Diseases of the Lung, Pleura and Mediastinum
Brief Title: Hyperspectral Imaging in Thoracic Surgery
Acronym: PILOT-Tx-HSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LungenClinic Grosshansdorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PILOT-Tx-HSI
Record Dates: First submitted 2021-02-25; First posted 2021-03-05 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2021-04

CONDITIONS: Bronchus Anastomosis; Bronchus Stump; Tissue Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HSI-Pilot (Experimental): Diagnostic hyperspectral imaging of the bronchus stump or bronchus anastomosis after lung resection and calculating the stump or anastomotic Perfusion measures, respectively
  Interventions: Device: HSI

INTERVENTIONS:
Device: HSI — diagnostic hyperspectral imaging

SUMMARY:
The aim of this study is to find out whether hyperspectral imaging enables bronchus stump and bronchus anastomosis oxygenation.

DETAILED DESCRIPTION:
The bronchus before lung resection and the bronchus stump or bronchus anastomosis, respectively, are investigated. The hyperspectral imaging camera head is placed and aligned over the surgical (camera and object distance: 30 cm for all measurements). The Field of view is illuminated by 8 halogen spots (20 W each) and 100 wavelengths in the wavelength range from 500 to 1000 nm were applied. The software calculates the tissue oxygenation [%] , organ-hemoglobin-index, near-infrared-Index and the tissue-water-index of the investigated tissue. The study was designed to investigate tissue oxygenation in the superficial (app. 1mm) and deeper layers (app. 4-6mm) of the bronchus before and after lung resection.

ELIGIBILITY:
Inclusion Criteria:

* lung resection or other resection via thoracotomy

Exclusion Criteria:

* Restriction of the ability to consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Oxygenation: Bronchus before lung resection | directly before lung resection
  Tissue perfusion of the bronchus before lung resection: Oxygenation (StO2) in %: Relative O2 saturation of the blood in superficial tissue layers (penetration depth: approx. 1 mm)
Oxygenation: Bronchus stump or bronchus anastomosis after lung resection | 10-15 minutes after lung resection
  Tissue perfusion of the bronchus stump or bronchus anastomosis after lung resection: Oxygenation (StO2) in %: Relative O2 saturation of the blood the in superficial tissue layers (penetration depth: approx. 1 mm)
Near Infrared Perfusion Index: Bronchus before lung resection | directly before lung resection
  Tissue perfusion of the bronchus before lung resection: Near Infrared Perfusion Index: Tissue perfusion in deeper tissue layers (penetration depth: 4-6mm)
Near Infrared Perfusion Index: Bronchus stump or bronchus anastomosis after lung resection | 10-15 minutes after lung resection
  Tissue perfusion of the bronchus stump or bronchus anastomosis after lung resection: Near Infrared Perfusion Index: Tissue perfusion in deeper tissue layers (penetration depth: 4-6mm)
Tissue-Hemoglobin index: Bronchus before lung resection | directly before lung resection
  Tissue perfusion of the bronchus before lung resection: Tissue-Hemoglobin index: Existing hemoglobin distribution in the tissue
Tissue-Hemoglobin index: Bronchus stump or bronchus anastomosis after lung resection | 10-15 minutes after lung resection
  Tissue perfusion of the bronchus stump or bronchus anastomosis after lung resection: Tissue-Hemoglobin index: Existing hemoglobin distribution in the tissue
Tissue-Water-Index: Bronchus before lung resection | directly before lung resection
  Tissue perfusion of the bronchus before lung resection: Tissue-Water-Index: Existing water distribution in the tissue
Tissue-Water-Index: Bronchus stump or bronchus anastomosis after lung resection | 10-15 minutes after lung resection
  Tissue perfusion of the bronchus stump or bronchus anastomosis after lung resection: Tissue-Water-Index: Existing water distribution in the tissue

CONTACTS AND LOCATIONS:
Overall Officials: David B. Ellebrecht, MD, Principal Investigator — LungenClinic Grosshansdorf
Locations (1):
- LungenClinic Großhansdorf, Großhansdorf, Germany

REFERENCES:
- [Derived] Ellebrecht DB, Kugler C. Intraoperative Determination of Bronchus Stump and Anastomosis Perfusion with Hyperspectral Imaging. Surg Innov. 2023 Jun;30(3):314-323. doi: 10.1177/15533506231157165. Epub 2023 Feb 21. PMID 36802983